CLINICAL TRIAL: NCT02798822
Title: Dental Arches Response to Haas-type RME Anchored to Deciduous vs Permanent Molars in Children With Unilateral Posterior Crossbite
Brief Title: Maxillary and Mandibular Arch Response to RME: a Multicentric Randomized Controlled Trial
Acronym: 6vsE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, ALESSANDRO UGOLINI, DDS MS PHD Researcher, University of Genova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80911110
Record Dates: First submitted 2013-08-02; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Posterior Crossbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RME on upper first permanent molars (Active Comparator): Intervention/Procedure: Rapid maxillary expansion. When RME was in situ, patients started the screw activation (Snap-lock expander screw, Forestadent, Pforzheim, Germany) of one-quarter turn a day (0.22 mm) until overcorrection was achieved (ie, the occlusal surface of the first maxillary palatal cusp contacted the occlusal surface of the mandibular first molar facial cusp), and the RME remained in place for 10 months. The screw was turned for 35 ± 6 days for Gr6, and the average treatment time was 12 ± 1.3 months.
  Interventions: Procedure: Rapid maxillary expansion
- RME on upper second deciduous molars (Active Comparator): Intervention/Procedure: Rapid maxillary expansion. When RME was in situ, patients started the screw activation (Snap-lock expander screw, Forestadent, Pforzheim, Germany) of one-quarter turn a day (0.22 mm) until overcorrection was achieved (ie, the occlusal surface of the first maxillary palatal cusp contacted the occlusal surface of the mandibular first molar facial cusp), and the RME remained in place for 10 months. The screw was turned for 41 ± 8 days, and the average treatment time was 12 ± 1.3 months.
  Interventions: Procedure: Rapid maxillary expansion

INTERVENTIONS:
Procedure: Rapid maxillary expansion — When rapid maxillary expander was in-situ, patients waited 7 days before starting the screw activation of one quarter turn a day (0.22 mm) until overcorrection. Expansion was considered adequate when the occlusal surface of the first maxillary palatal cusp contacted the occlusal surface of the mandibular first molar facial cusp. When was achieved, rapid maxillary expander stayed in place for 10 months.

SUMMARY:
Posterior crossbite is a common clinical condition often associated with transverse maxillary deficiency and functional mandibular shift. This frequent malocclusion is not self-correcting and can lead to the development of craniofacial asymmetries and mandibular dysfunction.

The aim of the current study was to evaluate maxillary and mandibular arch widths' response to RME when it is anchored to the upper second deciduous molars or to the upper first permanent molars and to create a decision-making protocol for RME therapy in mixed-dentition patients.

DETAILED DESCRIPTION:
The effects of rapid maxillary expansion (RME) on the maxillary complex have been highly investigated,4 reporting a maximum maxillary intermolar and intercanine width increase of 6.7 mm and 5.3 mm,5 respectively, when RME is banded on upper first permanent molars.

Literature also reported cases of periodontal and endodontic damage on RME anchoring teeth; therefore, some authors have suggested banding RME on primary teeth and reporting also different mean intermolar (3.6-4.1 mm) and intercanine width increases (5-5.9 mm).

Few studies have investigated the changes in molar dental tipping and inclinations (on average from 3° up to 16.7°) following RME but comprised difficult (ie, barium sulfate solution) and more invasive examinations such as computed tomography and cone beam computed tomography (CBCT) Few articles concerning the indirect effects on mandibular arch following RME reported a low but statistically significant increase of lower intermolar (0.66-0.97 mm) and intercanine width (0.9 mm). Since no studies in the literature have analyzed the differences in permanent vs primary molars as anchoring teeth for RME, the decision to band the permanent deciduous molars did not follow a clinical protocol, but an individual decision was made for each patient based on clinician experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients in mixed dentition
* Unilateral posterior crossbite at least of the first permanent molar
* Upper deciduous second molars available as RME anchoring teeth

Exclusion Criteria:

Primary exclusion criteria

* Previous orthodontic treatment
* Hypodontia in any quadrant excluding third molars
* Inadequate oral hygiene
* Temporomandibular joint disorders
* Craniofacial abnormalities
* Secondary exclusion criteria
* Lack of records
* Need for lingual arch
* Lack of consensus
* Need for other orthodontic treatment during rapid maxillary expansion

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Crossbite correction (binary outcome yes/no: clinical evaluation in vivo and on digital dental casts) | 5 months

SECONDARY OUTCOMES:
Crossbite correction stability (binary outcome yes/no: clinical evaluation in vivo and measured on digital dental casts) | 10 months
Canine angulation (degrees of transverse expansion measured on digital dental casts) | 5 months
Canine angulation (degrees of transverse expansion measured on digital dental casts) | 10 months
Molar angulation (degrees of transverse expansion measured on digital dental casts) | 5 months
Molar angulation (degrees of transverse expansion measured on digital dental casts) | 10 months
Molar expansion (mm of transverse expansion measured on digital dental casts) | 5 months
Molar expansion (mm of transverse expansion measured on digital dental casts) | 10 months
Canine Expansion (mm of transverse expansion measured on digital dental casts) | 5 months
Canine Expansion (mm of transverse expansion measured on digital dental casts) | 10 months
Upper and lower incisor angulation and rotation (changes in mm and degrees of dental angulation and rotation measured on digital dental casts and Dental digital X-ray) | 10 months

OTHER OUTCOMES:
Cephalometric evaluation of craniofacial growth (changes in mm and degrees of craniofacial skeletal growth measured on dental digital X-ray) | 10 months
Cephalometric evaluation of morphology of the cervical vertebrae (changes in mm and degrees of cervical vertebrae morphology on dental digital X-ray) | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Ugolini, DDS, PhD, Principal Investigator — University of Genova
Locations (3):
- Italy (3):
  - Ortohdontic Department - Univesity of Genoa, Genova
  - Ortohdontic Department - Univesity of Siena, Siena
  - Orthodontic Department - University of Varese, Varese

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cerruto C, Ugolini A, Di Vece L, Doldo T, Caprioglio A, Silvestrini-Biavati A. Cephalometric and dental arch changes to Haas-type rapid maxillary expander anchored to deciduous vs permanent molars: a multicenter, randomized controlled trial. J Orofac Orthop. 2017 Sep;78(5):385-393. doi: 10.1007/s00056-017-0092-2. Epub 2017 Apr 10. PMID 28397083